CLINICAL TRIAL: NCT02495064
Title: Mometasone Furoate Cream Reduces Acute Radiation Dermatitis in Head and Neck Squamous Cell Carcinomas' Patients Receiving Radiation Therapy
Brief Title: Mometasone Furoate Cream Reduces Acute Radiation Dermatitis in Head and Neck Squamous Cell Carcinomas' Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yao Liao (Other)
Responsible Party: Sponsor-Investigator, Yao Liao, Doctor of oncology department in Mianyang Central Hospital, Mianyang Central Hospital
Organization: Mianyang Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MianyangCH
Record Dates: First submitted 2015-01-25; First posted 2015-07-13 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Early Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mometasone Furoate Cream(MF) (Experimental): participants will be given conventional Chemoradiotherapy and MF.
  MF Brief introduction:
  Generic name :Mometasone Furoate Cream. Dosage form:Each gram of Mometasone Furoate Cream contains mometasone furoate, USP in a cream base of hexylene glycol, phosphoric acid, propylene glycol stearate, stearyl alcohol and ceteareth-20, titanium dioxide, aluminum starch octenylsuccinate, white wax, white petrolatum, and purified water.
  Dosage:Apply a thin film of Mometasone Furoate Cream to the affected skin areas once daily during radiotherapy.
  It is a corticosteroid indicated for the relief of the inflammatory and pruritic manifestations of corticosteroid-responsive dermatoses.
  Interventions: Drug: Mometasone Furoate Cream
- Chemoradiotherapy (No Intervention): conventional Chemoradiotherapy only

INTERVENTIONS:
Drug: Mometasone Furoate Cream — One side of patients' neck will begain to use MF cream from the first day of radiation therapy.
  Other Names: Eloson
  Arms: Mometasone Furoate Cream(MF)

SUMMARY:
Radiation dermatitis is an acute effect of radiation therapy,Especially in the neck skin of head and neck squamous cell carcinomas' patients.The investigators wanted to confirm the benefit of mometasone furoate (MF) in preventing acute radiation reactions, as shown in a previous study.

DETAILED DESCRIPTION:
A randomized,self-comparative controlled trial was undertaken comparing MF cream with no cream administered from the first day of treatment for 5-6 weeks to prevent radiation dermatitis of neck during radiation therapy to the head and neck squamous cell carcinomas' Patients.

One side of patients' neck will begin to use MF cream from the first day of radiation therapy, while the other side accept no preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* pathological diagnosis for head and neck squamous cell carcinomas and
* going to have radiotherapy.

Exclusion Criteria:

* pregnant,
* lactating women,
* infants,
* elderly people with atrophy skin,
* allergic constitution patients,
* the corresponding parts of 5 radiotherapy skin ulceration or infection and
* allergic patients to Mometasone Furoate Cream.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the mean Radiation Therapy Oncology Group (RTOG) skin dermatitis score | seven weeks
  The investigators descriph the skin dermatitis scores every week during radiation therapy and the later two weeks as follows:The scores were 0 = no visible change; 1 = faint or dull erythema; 2 = tender or bright erythema with or without moist desquamation; 3 = patchy moist desquamation with moderate edema; and 4= confluent moist desquamation with pitting edema.

CONTACTS AND LOCATIONS:
Overall Officials: Wang dong, Principal Investigator — Health Bureau of Mian Yang
Locations (1):
- oncology department of Mian yang central Hosptial, Mianyang, Sichuan, China